CLINICAL TRIAL: NCT00951093
Title: The Impact of Gastric Bypass on Gastroesophageal Reflux Disease in Patients With Morbid Obesity: a Prospective Study Based on Montreal Consensus
Brief Title: Gastroesophageal Reflux Disease (GERD) Before and After Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Clinica Gastrobese (Other)
Responsible Party: Principal Investigator, Carlos AS Madalosso, Director of Department of Metabolic and Bariatric Surgery, Clinica Gastrobese
Other Study IDs: GASTROBESE-004
Record Dates: First submitted 2009-08-02; First posted 2009-08-04 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disease; Morbid Obesity
Keywords: GERD; Gastric bypass
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients assessed for GERD: Patients who had an open gastric bypass were assessed for GERD before and after surgery following the Montreal Consensus through a validated questionnaire in Portuguese language
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Procedure: Gastric bypass — Open Silastic® ring Roux-en Y gastric bypass was performed through an upper midline incision. A gastric pouch was created by dividing the stomach with a 10-cm stapler from the lesser curvature (7 cm vertically from the cardia) to 1 cm to the left of the Hiss angle. The estimated volume of the gastric pouch was 20 to 30 ml that was banded with a 6.5 cm long Silastic® ring. A gastrojejunal anastomosis was performed with two-layers hand sewn absorbable suture over a 1.2 cm bougie distal to the ring, keeping an alimentary limb with 100 cm in length, and a biliopancreatic limb ranging 60 and 80 cm.

SUMMARY:
The hypothesis of this study was that gastric bypass (GBP) ameliorates gastroesophageal reflux disease (GERD) in morbidly obese patients.

DETAILED DESCRIPTION:
The investigators studied the impact of this surgical procedure on GERD in patients with morbid obesity.

Esophageal syndromes were evaluated according to the Montreal Consensus, where troublesome symptoms were defined as score ≥ 2 on a validated questionnaire of symptoms for Portuguese language along with esophageal syndromes with injury assessed through upper endoscopy.

Esophageal acid exposure was determined through 24h pH monitoring. Increased acid exposure was characterized when total esophageal pH < 4 for at least 4% of the total monitoring time.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity
* Acceptance to undergo open gastric bypass

Exclusion Criteria:

* Prior gastroesophageal surgery
* Achalasia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2007-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos AS Madalosso, PhD, Principal Investigator — Clinica Gastrobese
Locations (1):
- Clínica Gastrobese, Passo Fundo, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Madalosso CA, Gurski RR, Callegari-Jacques SM, Navarini D, Thiesen V, Fornari F. The impact of gastric bypass on gastroesophageal reflux disease in patients with morbid obesity: a prospective study based on the Montreal Consensus. Ann Surg. 2010 Feb;251(2):244-8. doi: 10.1097/SLA.0b013e3181bdff20. PMID 20010088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 126 consecutive patients were assessed on site (Gastrobese Clinic) between March and October 2007, 94 met the criteria.
  8 patients were lost to follow-up, 4 before and 4 after GBP. Out of those, 15 were lost to follow-up and 18 refused to follow through, resulting on the actual 53 patients.
Groups:
- Patients Assessed for GERD: Patients assessed for GERD before and after Gastric Bypass Surgery
Period: Before GBP
Arm/Group | Patients Assessed for GERD
Started | 53
Completed | 53
Not Completed | 0
Period: 6 Months After GBP
Arm/Group | Patients Assessed for GERD
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients were enrolled irrespective of GERD symptoms according to the following criteria:
  1. age between 18 and 70 years,
  2. BMI ≥ 40 kg/m2 or ≥ 35 kg/m2 combined with significant comorbidities,
  3. absence of gastroesophageal surgery, and
  4. consent to undergo open GBP
Groups:
- Patients Assessed for GERD: Patients who had an open gastric bypass were assessed for GERD before and after surgery.
Arm/Group | Patients Assessed for GERD
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.26 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 15
Region of Enrollment [Number; unit: participants]
  Brazil | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Presenting Reflux Symptoms
Description: Prevalence of typical reflux syndrome according to the Montreal Consensus. This Consensus institutes that GERD can be outlined when troublesome symptoms and/or complications induced by reflux of the gastric content back to the esophagus are present.
  In order to assess such troublesome symptoms a validated questionnaire translated into Portuguese language was used.
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Number; unit: participants
Groups:
- Before GBP: Patients assessed for GERD before Gastric Bypass Surgery
- 6 Months After GBP: Patients assessed for GERD 6 months after Gastric Bypass Surgery
- 39 Months After GBP: Patients assessed for GERD 39 months after Gastric Bypass Surgery
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
participants | 31 | 8 | 5
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p < 0.001, Friedman´s test — P value adjusted for multiple comparisons; followed by nonparametric pairwise multiple comparisons

2. Primary Outcome: Number of Participants With Esophageal Injury
Description: Syndromes with esophageal injury were represented exclusively by the presence of reflux esophagitis
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Number; unit: participants
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
participants | 24 | 17 | 10
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p = 0.002, Friedman´s test; followed by nonparametric pairwise multiple comparisons

3. Primary Outcome: Number of Participants With Gastroesophageal Reflux Disease (GERD)
Description: Prevalence of GERD in patients characterized according to troublesome symptomatic syndromes assessed through a validated questionnaire based on the Montreal Consensus.
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Number; unit: participants
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
participants | 34 | 21 | 12
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p < 0.001, Friedman´s test

4. Primary Outcome: Total Esophageal Acid Exposure at 24h pH Monitoring
Description: Esophageal acid exposure was measured through 24h pH monitoring. During the entire period, esophageal pH was measured and recorded as the percent of time pH was below 4.
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
percentage of time | 5.1 [2.3 to 8.0] | 1.2 [0.3 to 6.3] | 0.1 [0.0 to 1.4]
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p < 0.020, Wilcoxon (Mann-Whitney); followed by nonparametric pairwise multiple comparisons

5. Primary Outcome: Esophageal Acid Exposure at 24h pH Monitoring in Upright Position
Description: Esophageal acid exposure was measured through 24h pH monitoring. Esophageal pH was measured and recorded as the percent of time pH was below 4 while participant in upright position
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
percentage of time | 5.9 [3.6 to 8.7] | 0.8 [0.2 to 2.7] | 0.1 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); followed by nonparametric pairwise multiple comparisons

6. Primary Outcome: Esophageal Acid Exposure at 24h pH Monitoring in Supine Position
Description: Esophageal acid exposure was measured through 24h pH monitoring. Esophageal pH was measured and recorded as the percent of time pH was below 4 while participant in supine position
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
percentage of time | 1.8 [0.1 to 6.3] | 0.5 [0 to 10] | 0.0 [0.0 to 0.4]
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); followed by nonparametric pairwise multiple comparisons

7. Primary Outcome: Number of Participants With Increased Acid Exposure
Description: Increased Acid Exposure occurs when esophageal pH is <4 for a period longer than 4% of the total test time on a 24h pH monitoring.
Time Frame: Before GBP, 6 months after GBP and 39 months after GBP
Measure: Number; unit: participants
Arm/Group | Before GBP | 6 Months After GBP | 39 Months After GBP
Number analyzed (Participants) | 53 | 53 | 53
participants | 31 | 16 | 9
Statistical Analysis 1: Comparison: Before GBP vs 6 Months After GBP vs 39 Months After GBP; Test type: Superiority or Other; p < 0.001, Friedman´s test; followed by nonparametric pairwise multiple comparisons

ADVERSE EVENTS:
Description: Serious and Other Non-Serious Adverse Events were not collected/assessed during the study
Arm/Group | Patients Assessed for GERD
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes